CLINICAL TRIAL: NCT03936101
Title: Prenatal Genetic Diagnosis by Genomic Sequencing: A Prospective Evaluation
Brief Title: Prenatal Genetic Diagnosis by Genomic Sequencing
Acronym: PrenatalSEQ
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Baylor College of Medicine (Other); University of North Carolina (Other); The George Washington University Biostatistics Center (Other); Oregon Health and Science University (Other); Children's Hospital Medical Center, Cincinnati (Other); The University of Texas Health Science Center, Houston (Other); Broad Institute of MIT and Harvard (Other); The Jackson Laboratory (Other)
Responsible Party: Principal Investigator, Ronald J Wapner, MD, Director, Reproductive Genetics, Department of OBGYN, Columbia University
Other Study IDs: AAAS2118; R01HD055651 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-05-03 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Fetal Structural Anomalies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Remaining DNA from trios will be stored in a biorepository. Plasma from Streck tubes will be retained as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prenatally Sequenced Group: 750 trios with fetal structural anomalies who receive prenatal sequencing from the study
  Interventions: Diagnostic Test: Prenatal Genomic Sequencing
- No Prenatal Sequencing (Unsequenced) Group: 350 trios with fetal structural anomalies who do not have prenatal sequencing

INTERVENTIONS:
Diagnostic Test: Prenatal Genomic Sequencing — Whole genome sequencing (which initially will be masked and reported as exome only)
  Groups: Prenatally Sequenced Group

SUMMARY:
This study is evaluating the impact of prenatal sequencing on the management of fetuses with ultrasound abnormalities. The hypothesis is that a significant subset of fetal abnormalities have a genetic cause that can be identified by sequencing and that prenatal knowledge of this information will improve prenatal care, reduce unnecessary diagnostic testing, reduce the cost of care, and improve the quality of life for both the child and the family.

DETAILED DESCRIPTION:
Whole exome and whole genome sequencing (WGS) have expanded the ability to determine the genetic etiology of previously undiagnosed disorders. This study is a multicenter prospective cohort study to evaluate the emerging technology of sequencing for the management of fetuses with structural anomalies. The hypothesis is that a significant subset of fetal structural anomalies has a genetic etiology identifiable by sequencing and that prenatal knowledge of this information will improve perinatal care, reduce unnecessary diagnostic testing, reduce the cost of care, and improve quality of life for both the child and the family. The aims of this study are to investigate these multiple aspects of prenatal sequencing in a single study with an innovative integrated prospective design, which will permit a robust evaluation of the benefits and risks of delivering diagnostic and prognostic genetic testing results in a prenatal setting.

The study will determine, in a sequential population of pregnancies with selected fetal structural anomalies and a negative or non-causal chromosomal microarray (CMA), the frequency of pathogenic, likely pathogenic, and uncertain genomic variants identifiable by sequencing. To determine the impact of this information on clinical care, a control population of unsequenced pregnancies with similar structural anomalies will be prospectively recruited and the infants from both cohorts will be followed up to 1 year of age. This study component will evaluate differences in healthcare management and cost through discharge from hospital post-delivery, and perinatal and infant outcomes through 1 year of life. The educational, counseling and psychosocial impact of sequencing results during the prenatal period, in the nursery and through 1 year of life also will be evaluated. Since the analytical and clinical tools needed for the full translation of sequencing into care are still developing, optimization of bioinformatic tools to improve identification of pathogenic and likely pathogenic mutations associated with prenatal phenotypes of established disease genes will be investigated, as well as identification of new genes associated with presently undiagnosed fetal/neonatal phenotypes. This study will provide an in-depth evaluation of the prenatal diagnostic value of sequencing prior to its responsible introduction into practice and will provide independent data to guide its translation.

ELIGIBILITY:
Inclusion Criteria:

Prenatal sequencing group

1. Fetus identified by ultrasound and/or MRI with at least one of the following:

   1. One or more major structural anomalies (Appendix A)
   2. A nuchal translucency measurement of ≥ 3.5 mm
   3. A fetus less than 24 weeks 0 days gestation with normal anatomy and sonographically estimated fetal weight <5th %ile without maternal hypertension, type I diabetes, or other maternal disorders known to alter fetal growth.
2. Negative prenatal CMA (or those with CMA findings not related to the ultrasound finding)
3. Singleton or twin gestation
4. Gestational age less than 36 weeks, 0 days to allow for availability of sequencing results before delivery

Unsequenced Group

1. Fetus identified by ultrasound and/or MRI with at least one of the following:

   1. One or more major structural anomalies (Appendix A)
   2. A nuchal translucency measurement of ≥ 3.5 mm
   3. A fetus less than 24 weeks 0 days gestation with normal anatomy and sonographically estimated fetal weight <5th %ile without maternal hypertension, type I diabetes, or other maternal disorders known to alter fetal growth
2. Negative prenatal or postnatal CMA (or those with CMA findings not related to the ultrasound finding)
3. Declined prenatal sequencing
4. Singleton gestation

Exclusion Criteria:

Prenatal Sequencing Group

1. Prenatal sequencing or planned prenatal sequencing performed outside of the study, including gene panels
2. Maternal or paternal age less than 18 years old
3. Proven infectious or teratogenic cause of fetal anomaly
4. Planned termination of the pregnancy
5. Unavailable blood or saliva samples from both biologic parents prior to sequencing
6. Parental unwillingness to participate in 1 year postnatal follow-up
7. Language barrier (non-English or Spanish speaking)
8. Previous consent to the unsequenced prenatal group or enrollment in a previous pregnancy

Unsequenced Group

1. Maternal or paternal age less than 18 years old
2. Proven infectious or teratogenic cause of fetal anomaly
3. Positive prenatal NIPT screening for trisomy 21,18 or 13. Positive 22q11.2 prenatal NIPT testing with consistent ultrasound findings is also an exclusion.
4. Planned termination of the pregnancy
5. Parental unwillingness to participate in 1 year postnatal follow-up
6. Language barrier (non-English or Spanish speaking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 1,100 pregnancies with fetal structural anomalies and meeting eligibility criteria will be enrolled into the study. Of these, 750 will undergo prenatal genomic sequencing (prenatal sequencing group) and the remaining 350 pregnancies will not have any prenatal genomic sequencing (unsequenced prenatal group).
  Enrollment of pregnancies with an isolated nuchal translucency measurements ≥ 3.5 mm will be restricted to 5% within each group (sequenced and unsequenced) and isolated estimated fetal weight <5th %ile also will be restricted to 5% for each group (sequenced and unsequenced).
Sampling Method: Non-Probability Sample
Enrollment: 1097 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (5):
- United States (5):
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital, Cincinnati Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas
  - UT Health Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH Genomic Data Sharing policy, sequencing data (including VCF files) and clinical data will be shared with other scientific investigators and through the controlled access dbGAP repository or comparable genomics commons, the Sequence Read Archive, and any NIH Birth Defects Commons that is established. A final dataset containing clinical and phenotypic data will be submitted to the NICHD data repository (DASH). In addition, new algorithms and allele frequency data will be shared with the newly developed Precision FDA platform as applicable.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study completion.
Access Criteria: Through dbGaP or other controlled access databases.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Signed informed consent was obtained from the mother and the genetic father of the fetus prior to any study procedures for prospective enrollment. Enrollment of participants in the retrospective unsequenced prenatal group occurred under a waiver of consent. The "participants" in this record refer to the fetuses from which all study data was collected.
Groups:
- Prenatally Sequenced Group: Pregnancies with fetal structural anomalies will undergo prenatal genomic sequencing.
- No Prenatal Sequencing (Unsequenced) Group: Pregnancies will not have any prenatal genomic sequencing.
Period: Overall Study
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Started | 751 | 346
Completed | 751 | 346
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group | Total
Number analyzed (Participants) | 751 | 346 | 1097
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Gestational age at diagnosis
  weeks | 20.4 [18.4 to 22.9] | 22.1 [20.0 to 25.4] | 21.0 [19.0 to 23.6]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex/gender was not collected from any fetus
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Maternal race/ethnicity: Black | 66 | 55 | 121
  Maternal race/ethnicity: White | 448 | 173 | 621
  Maternal race/ethnicity: Hispanic | 156 | 96 | 252
  Maternal race/ethnicity: Other | 81 | 22 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Of the 346 enrolled in the unsequenced comparison cohort, 150 were enrolled prospectively and 196 were retrospectively enrolled. Paternal race/ethnicity was not collected from the retrospective cohort.
  Paternal race/ethnicity was not collected from one participant in the sequenced arm.
  Participants
    Paternal race/ethnicity: number analyzed (Participants) | 750 | 150 | 900
    Paternal race/ethnicity: Black | 68 | 20 | 88
    Paternal race/ethnicity: White | 456 | 91 | 547
    Paternal race/ethnicity: Hispanic | 151 | 32 | 183
    Paternal race/ethnicity: Other | 75 | 7 | 82
Region of Enrollment [Number; unit: participants]
  United States | 751 | 346 | 1097
Anomaly systems involved [Count of Participants; unit: Participants]
  Single anomaly system | 474 | 234 | 708
  Multiple anomaly systems | 277 | 112 | 389
Type of anomaly [Count of Participants; unit: Participants]
  Cardiovascular | 193 | 150 | 343
  central nervous system | 203 | 79 | 282
  Craniofacial | 96 | 34 | 130
  Cystic hygroma (nuchal translucency (NT) ≥ 4.5 mm) | 74 | 4 | 78
  Effusion | 88 | 30 | 118
  Fetal growth restriction < 5th percentile | 65 | 26 | 91
  Gastro-intestinal tract | 90 | 46 | 136
  Genitourinary | 152 | 65 | 217
  NT ≥ 3.5 mm to < 4.5 mm without evidence of cystic hygroma | 31 | 3 | 34
  Osteoarticular | 164 | 69 | 233
  Intrathoracic | 66 | 44 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Reportable Variants
Description: Reportable variants: defined as either Pathogenic / Likely pathogenic (P/LP) or variant of uncertain significance (VUS) identified by sequencing and deemed reportable by the Variant Adjudication Committee.
Time Frame: At end of study, approx 4 years
Population: Only participants in the sequenced group were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
Participants
  P/LP | 114
  VUS | 22

2. Primary Outcome: Healthcare Costs
Description: Healthcare costs from time of diagnosis of anomaly to infant discharge between sequenced and unsequenced groups.
Time Frame: From time of diagnosis of anomaly to infant discharge
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 444 | 312
US dollars | 149985 (375687) | 165192 (350000)

3. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age of newborn at delivery (in weeks)
Time Frame: At time of delivery
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 751 | 346
weeks | 37.4 [35.0 to 39.0] | 38.0 [36.9 to 39.0]

4. Secondary Outcome: Neonatal Outcomes
Description: Neonatal outcomes will be compared and outcomes will be measured by the number of newborns who experience: need for ventilator support, sepsis, need for pressor support, need for extracorporeal membrane oxygenation (ECMO), metabolic abnormalities (e.g., acidosis, elevated uric acid, hypo-/hyperglycemia), intraventricular hemorrhage, periventricular leukomalacia, encephalopathy, and seizure.
Time Frame: Up to 28 days after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 751 | 346
Participants
  Mechanical ventilation | 222 | 151
  ECMO | 24 | 19
  Pressor support | 89 | 69
  Sepsis | 92 | 66
  Metabolic abnormalities | 192 | 91
  Intraventricular hemorrhage | 42 | 33
  Periventricular leukomalacia | 5 | 4
  Encephalopathy | 24 | 8
  Seizure | 20 | 16

5. Secondary Outcome: Number of Deaths
Description: Neonatal/infant death at time of discharge and at 12 months of age.
Time Frame: From discharge to 12 months postpartum
Measure: Number; unit: deaths
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 751 | 346
deaths | 75 | 37

6. Secondary Outcome: NICU Stay Duration
Description: Length of initial NICU stay and number of days spent in the hospital between initial discharge and 12 months of age.
Time Frame: From discharge to 12 months postpartum
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 751 | 346
days | 6.0 [0.00 to 29.0] | 11.0 [1.0 to 35.0]

7. Secondary Outcome: Length in Centimeters
Description: Infant length at 12 months of age.
Time Frame: 12 months postpartum
Population: Data was collected from participants who had a follow-up visit at 12 months postpartum.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 202 | 50
cm | 73.7 (6.3) | 73.6 (6.1)

8. Secondary Outcome: Weight in Kilograms
Description: Infant weight at 12 months of age.
Time Frame: 12 months postpartum
Population: Data was collected from participants who had a follow-up visit at 12 months postpartum.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 230 | 57
kg | 9.3 (1.5) | 9.6 (1.3)

9. Secondary Outcome: Score on Development by Ages and Stages Questionnaire (ASQ-3)
Description: Developmental outcomes defined by the following parameters: communication, gross motor, fine motor, problem solving and personal-social, at 12 months of age using ASQ-3. Lower scores are associated with developmental delay. For each developmental area, parents may answer YES=10, SOMETIMES=5, or NOT YET=0 by filling in a bubble for each item response. The full score range for each domain is 0 to 60.
  Cutoffs for each domain are: Communication 15.64, Gross Motor 21.49, Fine Motor 34.5, Problem Solving 27.32, Personal-Social 21.73
Time Frame: 12 months postpartum
Population: Only includes participants who completed the follow-up questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 152 | 38
score on a scale
  Communication | 45 [30 to 55] | 45 [30 to 55]
  Gross motor | 40 [15 to 60] | 43 [10 to 60]
  Fine motor | 50 [40 to 55] | 48 [35 to 55]
  Problem solving | 50 [35 to 55] | 45 [35 to 55]
  Personal-social | 45 [35 to 55] | 50 [35 to 55]

10. Secondary Outcome: Anxiety by Self-report Questionnaire
Description: Anxiety following result disclosure (or 8 weeks post enrollment for the unsequenced group), neonatal discharge and 12 months postpartum. The full score range is 0 to 21, where lower numbers represent lower anxiety (better outcome).
Time Frame: 2 weeks after disclosure of study sequencing results or 4 weeks after enrollment for the unsequenced group; 1 month after discharge from the hospital or end of the pregnancy if there was a fetal demise or pregnancy termination; 12-15 months postpartum
Population: Only includes participants who completed the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 672 | 143
score on a scale
  2 weeks after disclosure of sequencing results or 4 weeks after enrollment for the unsequenced group: number analyzed (Participants) | 468 | 84
  2 weeks after disclosure of sequencing results or 4 weeks after enrollment for the unsequenced group | 2.0 [1.0 to 5.5] | 3.0 [1.0 to 6.5]
  1 month after discharge from the hospital or end of the pregnancy | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 5.0]
  12-15 months postpartum: number analyzed (Participants) | 593 | 126
  12-15 months postpartum | 2.0 [0.0 to 5.0] | 2.0 [0.0 to 5.0]

11. Secondary Outcome: Depression by Self-report Questionnaire
Description: Depression following result disclosure (or 8 weeks post enrollment for the unsequenced group), neonatal discharge and 12 months postpartum. The full score range is 0 to 24, where a lower score represents lower depression (better outcome).
Time Frame: as for outcome 10
Population: Only includes participants who completed the questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
Number analyzed (Participants) | 674 | 142
score on a scale
  2 weeks after disclosure of sequencing results or 4 weeks after enrollment for the unsequenced group: number analyzed (Participants) | 474 | 83
  2 weeks after disclosure of sequencing results or 4 weeks after enrollment for the unsequenced group | 4.0 [1.0 to 8.0] | 5.0 [2.0 to 9.0]
  1 month after discharge from the hospital or end of the pregnancy | 4.0 [1.0 to 7.0] | 4.0 [1.0 to 8.0]
  12-15 months postpartum: number analyzed (Participants) | 593 | 128
  12-15 months postpartum | 3.0 [1.0 to 7.0] | 3.5 [1.0 to 7.0]

12. Secondary Outcome: Quality of Life by Self-report Questionnaire
Description: Quality of life for the patient and family at 12 months postpartum.
Time Frame: Approximately 4.5 years
Reporting Status: Not Posted, anticipated posting 2026-07

13. Secondary Outcome: QALY, Measured in Cost Per Year
Description: Incremental cost per Quality Adjusted Life Year (QALY).
Time Frame: Approximately 4.5 years
Reporting Status: Not Posted, anticipated posting 2026-07

14. Secondary Outcome: Total Number of Identified Phenotypes Associated With Disease- Sequenced Group ONLY
Description: Phenotypic Expansion: Apparent prenatal phenotypic expansion from currently defined pediatric phenotypes.
Time Frame: 12 months postpartum
Population: This outcome was only intended to be measured in participants in the Sequenced arm, as outlined in the study protocol. Data for this outcome was not collected from any participant in the Unsequenced arm.
Measure: Number; unit: phenotypes
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
phenotypes | 22

15. Secondary Outcome: Number of Participants With VUS - Sequenced Group ONLY
Description: Variants of uncertain significance (VUS) that have not yet been associated with this disease phenotype.
  This outcome was only intended to be measured in participants in the Sequenced arm, as outlined in the study protocol. Data for this outcome was not collected from any participant in the Unsequenced arm.
Time Frame: 12 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
Participants | 7

16. Secondary Outcome: Number of Participants With Variants Classified as GUS - Sequenced Group ONLY
Description: VUS subclassified as compelling variants in novel genes that are not yet disease associated (genes of uncertain clinical significance; GUS).
  This outcome was only intended to be measured in participants in the Sequenced arm, as outlined in the study protocol. Data for this outcome was not collected from any participant in the Unsequenced arm.
Time Frame: 12 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
Participants | 0

17. Secondary Outcome: Digital WES - Comparison of Coding and Non-coding Results - Sequenced Group ONLY
Description: Pathogenic, likely pathogenic and VUS variants identified by sequencing (coding and non-coding regions) compared with coding regions only (digital WES).
Time Frame: Approximately 4.5 years
Reporting Status: Not Posted, anticipated posting 2026-07

18. Secondary Outcome: Proband Only Versus Trio - Comparison of Results Between Trio and Proband Only - Sequenced Group ONLY
Description: Pathogenic, likely pathogenic and VUS variants identified by analysis of a proband alone compared to a proband-parent trio.
Time Frame: Approximately 4.5 years
Reporting Status: Not Posted, anticipated posting 2026-07

19. Secondary Outcome: Change in Management (Healthcare) as Determined by NICU Physician and Record Review - Sequenced Group ONLY
Description: Number of participants who had a change in management decisions attributable to genomic results, defined as changes to the patient's treatment plan or changes to the counseling of the patient/family regarding the immediate or long-term medical management.
  This outcome was only intended to be measured in participants in the Sequenced arm, as outlined in the study protocol. Data for this outcome was not collected from any participant in the Unsequenced arm.
Time Frame: From delivery until discharge or death (neonatal)
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
Participants | 72

20. Secondary Outcome: Parental Support Needs by Self-report Questionnaire - Sequenced Group ONLY
Description: Assessment of educational/counseling and social support needs of the mother and father. The full score range is 12 to 60, where a higher score represents a higher satisfaction with the experience (better outcome).
Time Frame: At sequencing completion, approximately 4.5 years
Population: Only includes participants in the sequenced group who completed the questionnaire
Measure: Median (Full Range); unit: score on a scale
Groups:
- Reported Variants: Participants in the Sequenced group who had reportable variants: defined as either Pathogenic / Likely pathogenic (P/LP) or variant of uncertain significance (VUS) identified by sequencing and deemed reportable by the Variant Adjudication Committee.
- No Reported Variants: Participants in the Sequenced group who did not have reportable variants.
Arm/Group | Reported Variants | No Reported Variants
Number analyzed (Participants) | 63 | 428
score on a scale | 56 [52 to 58] | 56 [51 to 60]

21. Secondary Outcome: Parental Understanding by Self-report Questionnaire - Sequenced Group ONLY
Description: Accuracy of parental understanding of genetic test results. The parental responses to the question "How well do you understand your prenatal genetic test results?" will be collected. All possible responses are: "Not at all", "A little bit", "Moderately", "Quite a bit", and "Extremely"
Time Frame: At sequencing completion, approximately 4.5 years
Population: Only includes participants in the sequenced group who completed the questionnaire
Measure: Number; unit: parental responses
Arm/Group | Reported Variants | No Reported Variants
Number analyzed (Participants) | 67 | 458
parental responses
  Not at all | 0 | 3
  A little bit | 1 | 22
  Moderately | 5 | 83
  Quite a bit | 43 | 205
  Extremely | 18 | 145

22. Secondary Outcome: Number of Participants Who Had a Change in the Sequencing Result - Sequenced Group ONLY
Description: Reinterpretations of sequencing results that lead to a change in classification of sequencing variants.
  This outcome was only intended to be measured in participants in the Sequenced arm, as outlined in the study protocol. Data for this outcome was not collected from any participant in the Unsequenced arm.
Time Frame: From sequencing completion to data analysis period, up to 4.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
Participants | 7

23. Secondary Outcome: Turnaround Time - Sequenced Group ONLY
Description: Turnaround time of sequencing components and how it changes over time. This outcome was only intended to be measured in participants in the Sequenced arm, as outlined in the study protocol. Data for this outcome was not collected from any participant in the Unsequenced arm.
Time Frame: Time from sequencing initiation until study site result, up to 38 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prenatally Sequenced Group
Number analyzed (Participants) | 751
days | 11.5 (5.4)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 months
Arm/Group | Prenatally Sequenced Group | No Prenatal Sequencing (Unsequenced) Group
All-Cause Mortality (participants affected / at risk) | 75/751 | 37/346
Serious Adverse Events (participants affected / at risk) | 0/751 | 0/346
Other Adverse Events (participants affected / at risk) | 0/751 | 0/346

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT03936101/Prot_SAP_000.pdf